CLINICAL TRIAL: NCT00496535
Title: A Phase I/II Safety, Tolerability, and "Proof of Concept" Study of TNFerade™ Biologic in Combination With Concomitant Radiotherapy, Fluorouracil, and Hydroxyurea (TNF-FHX) for Patients With Unresectable Recurrent Head and Neck Cancer
Brief Title: A Study of TNFerade™ Biologic With Concomitant Radiotherapy, Fluorouracil, and Hydroxyurea (TNF-FHX) in Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GenVec (Industry)
Responsible Party: Paul Fischer, PhD, GenVec
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GV-001.011; GV-001.011 (TNF-CORE)
Record Dates: First submitted 2007-07-02; First posted 2007-07-04 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2011-05

CONDITIONS: Head and Neck Cancer; Head and Neck Neoplasms
Keywords: head; neck; cancer; neoplasm
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms

INTERVENTIONS:
Drug: TNFerade biologic

SUMMARY:
The primary objective of the first phase is to determine the safety, the maximum tolerated dose (MTD) and dose-limiting toxicity of TNFerade in combination with the previously studied combination of Fluorouracil (5FU), Hydroxyurea (HU) and standard daily radiotherapy in patients with recurrent head and neck cancer (RHNC). All chemoradiotherapy is administered on a "week-on/week-off" schedule. The primary objective of the second phase II is to determine the locoregional control rate at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer
* Patients must have a locoregional tumor amenable to reirradiation with curative intent.
* disease, or the majority of disease, should be accessible to injection via direct intratumoral injection
* Life expectancy of greater than 12 weeks
* Age > 18 years
* ECOG performance status 0-1

Exclusion Criteria:

* Metastatic disease
* History of malignancy (other than head and neck cancer) in the last 2 years except carcinoma in situ of the cervix or bladder, non-melanomatous skin cancer, or localized early stage prostate cancer, with patients continually disease free, or cancers that are not felt to influence treatment for head and neck cancer and life expectancy of patient
* Patients may not be receiving any other investigational agents currently or within the 4 weeks prior to study Day 1
* Active infection of any type
* Chronic treatment for greater than 6 months with steroids
* Pregnant or lactating women
* Patients with known history of cerebral vascular disease; stroke or TIA within the last 6 months
* Patients with history of documented thrombosis (PE or DVT), or known coagulopathy or thrombophilia, or evidence of DVT / thromboembolic event upon enrollment
* Patients receiving hormone replacement therapy or hormonal contraceptives within two weeks of day 1
* Patients who have undergone surgery within the last 1 month prior to day 1
* Patients with active carotid artery involvement or status post carotid artery graft / stenting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
locoregional control at 24 months

SECONDARY OUTCOMES:
Locoregional control at 3, 6 and 12 months, as well as tumor response rate, progression-free survival at 3, 6, 12 and 24 months, and the rate of metastases at 3, 6, 12 and 24 months will also be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Everett Vokes, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- University of Chicago, Chicago, Illinois, United States